CLINICAL TRIAL: NCT05987618
Title: Oral Appliances With and Without Elastic Bands to Treat Obstructive Sleep Apnea: A Randomized Crossover Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REKVEST550079
Record Dates: First submitted 2023-03-06; First posted 2023-08-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Sleep Apnea, Obstructive
Keywords: oral appliance; elastic bands
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The technician scoring the sleep recordings investigating the objective effect of oral appliance treatment with or without elastic bands, will be blinded to which treatment modality the patients are using.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral appliance with elastic bands (Experimental): Oral appliance therapy with elastic bands.
  Interventions: Device: Oral appliance with elastic bands
- Oral appliance without elastic bands (Active Comparator): Oral appliance therapy without elastic bands.
  Interventions: Device: Oral appliance without elastic bands

INTERVENTIONS:
Device: Oral appliance with elastic bands — The elastic bands are attached to hooks on both the upper and lower appliance, and on both sides. The elastic bands will be carefully selected not to interfere with retention of the oral appliance. The strongest elastic bands that do not interfere with retention of the oral appliance will be chosen, probably within the range of 85-170 grams (3/8" - 3/16").
  Other Names: Masel Geoshapes elastomerics
  Arms: Oral appliance with elastic bands
Device: Oral appliance without elastic bands — The oral appliance without the elastic bands.
  Arms: Oral appliance without elastic bands

SUMMARY:
The goal of this randomized crossover trial is to investigate the effect of elastic bands attached to oral appliances to minimize mouth opening during sleep in obstructive sleep apnea (OSA) patients. The main questions it aims to answer are:

* Are the success rates (>50% reduction of AHI) of oral appliances with elastic bands superior to oral appliances treatment without elastic bands in treatment of moderate and severe OSA?
* Are there predictors that can identify patients that will benefit from use of elastic bands in oral appliance treatment of OSA?
* Are there predictors that can identify patients that are classified as non-responders to oral appliance treatment in general, both with and without elastic bands?

Participants will be treated with oral appliances with and without elastic bands for 3 weeks, in randomized order. At the end of each 3-week period, the effect of the treatment will be investigated with sleep registrations and questionnaires.

After the completion of both 3-week periodes, patients will continue using their preferred treatment modality (with or without elastic bands) and the oral appliance will be titrated if suboptimal treatment effect.

DETAILED DESCRIPTION:
69 patients with moderate or severe OSA referred to Center of Sleep Medicine, Haukeland University Hospital (HUS), for oral appliance treatment will be invited to participate in the study.

The oral appliances will be produced with 63% and 69% of maximal protrusion for patients with moderate and severe OSA, respectively. Patients will be randomized to treatment with or without elastic bands before the oral appliance is fitted to the patient.

3 weeks after delivery, the subjective and objective effect of the treatment are investigated with questionnaires and home sleep testing with polygraphic sleep apnea recordings. The sleep recordings will be manually scored using scoring rules in accordance with the 2012 AASM guidelines. All sleep recording will be scored by the sane technician blinded to the treatment modality (with or without elastics).

Following, the patients will change treatment modality (with or without elastics), with identical investigation of objective and subjective treatment effect after 3 weeks of treatment.

If patients are not able to use their oral appliance due to side effects/discomfort at any point during the 3 week period, the issues are handled adequately, and control of the treatment is postponed for 2 week if remaining time to the planned control is <2 weeks. Patients are encouraged to make contact if side effects/discomfort related to the treatment are experienced.

After both treatment modalities (with and without elastic bands) are tested for 3 weeks, patients choose what treatment modality they want to continue treatment using, based on adherence, objective and subjective treatment effect. Treating physician will advice patients to choose the treatment that reduced their apnea-hypopnea index the most.

Objective treatment outcomes are classified following established success criteria:

* Success criterion 1: AHI < 5
* Success criterion 2: AHI < 10 and > 50% reduction of baseline AHI
* Success criterion 3: ≥50% reduction of baseline AHI
* Failure: <50% reduction of AHI from baseline

If success criterion 1 or 2 is not reached using the preferred treatment modality during the initial 3 week period, the oral appliance is titrated until it considered optimal. Following, the objective and subjective effect of the treatment is investigated with questionnaires and sleep recordings similar to initial treatment.

The patients with persistent <50% reduction of AHI from baseline after the oral appliance is optimally titrated will be offered treatment with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe OSA
* Non-compliant and/or non-responder to CPAP-treatment
* Considered for treatment with Somnodent Fusion (second line oral appliance - indicated when retention on remaining teeth is insufficient to retain Narval CC)
* Participate in the "Sleep registry" at Center for Sleep Medicine, Haukeland University Hospital

Exclusion Criteria:

* Mild OSA or no OSA
* Considered for treatment with Narval CC (first line oral appliance)
* Patients with insufficient amount of teeth to retain an oral appliance
* Patients with full denture
* Patients that do not speak and/or read Norwegian language
* Patients that are not competent to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Difference in success (>50% reduction in AHI) of oral appliance treatment with and without elastic bands. | The difference in success is investigated using PG-measures from controls 3 and 6 weeks after treatment start, at the end of the period with 3 weeks of oral appliance treatment with and without elastic bands.
  The objective effect of the treatment will be measured using ambulatory polypgrahic examination (PG) with a type IV device (Nox T3).

SECONDARY OUTCOMES:
Difference in reported compliance with oral appliance treatment with and without elastic bands. | The difference in reported compliance will be measured using data from controls 3 and 6 weeks after treatment start, at the end of the period with 3 weeks of oral appliance treatment with and without elastic bands.
  Compliance with oral appliance treatment both with and without elastic bands will be reported through questionnaires regarding average usage per night measured in hours, and average usage per week measured in number of nights.
Difference in reported side effects with oral appliance treatment with and without elastic bands. | The difference in reported side effects will be measured using data from controls 3 and 6 weeks after treatment start, at the end of the period with 3 weeks of oral appliance treatment with and without elastic bands.
  Side effects from oral appliance treatment both with and without elastic bands will be reported through questionnaires.
Difference in reported symptoms of anxiety and depression following oral appliance treatment with and without elastic bands. | Symptoms of anxiety and depression following oral appliance treatment will be measured using data from controls 3 and 6 weeks after treatment start, at the end of the period with 3 weeks of oral appliance treatment with and without elastic bands.
  Symptoms of anxiety and depression following oral appliance treatment both with and without elastic bands will be reported through questionnaire, using the Hospital Anxiety and Depression Scale.
Difference in subjective reported effect of oral appliance treatment with and without elastic bands. | The difference in subjective effect is investigated using the questionnaires from controls 3 and 6 weeks after treatment start, at the end of the period with 3 weeks of oral appliance treatment with and without elastic bands.
  Subjective effect of the treatment will be measured using questionnaires regarding effect on daytime somnolence, snoring, quality of life, and effect on bed side partners experienced quality of sleep.
Difference in reported insomnia and fatigue following oral appliance treatment with and without elastic bands. | The difference is investigated using the questionnaires from controls 3 and 6 weeks after treatment start, at the end of the period with 3 weeks of oral appliance treatment with and without elastic bands.
  Reported insomnia and fatigue following oral appliance treatment will be measured using questionnaires.
Variables associated with success of oral appliance treatment with elastic bands. | The variables included in the analysis will be extracted from controls 3 and 6 weeks after treatment start, at the end of the period with 3 weeks of oral appliance treatment with and without elastic bands.
  Both objective and subjective variables will be investigated to see if they may be associated with success with oral appliance treatment with elastic bands. This may better the selection of which patients are recommended oral appliance treatment with elastic bands. The objective variables investigated will be variables from the PG-examination (AHI, ODI, AHI supine, time in supine position, time <90% SaO2, average SaO2), measures of jaw function and occlusal characteristics (overjet, overbite, max protrusion, max mouth opening, angle class), and TMD-variables. Subjective variables will mainly be investigated to see if there are associations with adherence to oral appliance treatment with elastic bands. Patients will fill out a questionnaire regarding how different variables affect their choice of treatment (oral appliance with or without elastics). Variables included in the questionnaire will be objective effect, subjective effect, comfort and manageability.
Variables affecting choice of treatment after completed trial period (oral appliance with or without elastic bands) | Variables affecting choice of treatment after completed trial period will be collected after the two 3-week periodes of using oral appliance with and without elastic bands are completed.
  Following two 3-week periods of oral appliance treatment with and without elastic bands in randomized order, the patients will choose whether they wish to continue oral appliance treatment with or without elastic bands. They will be asked to justify their choice of treatment using a questionnaire, where they will be asked to grade in what degree different variables affected their choice of treatment.
Variables associated with success of oral appliance treatment. | The variables included in the analysis will be extracted from the final control after the oral appliance is considered optimally titrated. This may be after 6 weeks, but if suboptimal effect, it may be from final control >9 weeks after treatment start.
  Both objective and subjective variables will be investigated to see if they may be associated with success with oral appliance treatment in general. The objective variables investigated will be variables from the PG-examination (AHI, ODI, AHI supine, time in supine position, time <90% SaO2, average SaO2), measures of jaw function and occlusal characteristics (overjet, overbite, max protrusion, max mouth opening, angle class), and TMD-variables. Subjective variables will mainly be investigated to see if there are associations with adherence to oral appliance treatment. The associations between above mentioned variables and success with oral appliance treatment will be investigated, as well as the association between the variables and adherence to oral appliance treatment and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Johansson, PhD, Principal Investigator — University of Bergen
Locations (1):
- Center of Sleep Medicine, Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Derived] Opsahl UL, Berge M, Lehmann S, Bjorvatn B, Johansson A. Prediction of non-responders to oral appliance treatment of obstructive sleep apnea: a pilot study. Sleep Breath. 2025 Apr 15;29(2):159. doi: 10.1007/s11325-025-03315-1. PMID 40232353